CLINICAL TRIAL: NCT01976260
Title: A Pilot, Split-Face Randomized, Evaluator Blinded Study on the Effectiveness of a Bipolar Fractional Radiofrequency System Versus 1550-nm Fractional Photothermolysis for the Treatment of Acne Scars.
Brief Title: A Pilot Study Testing Fractional Radiofrequency Versus Fractional Photothermolysis for the Treatment of Acne Scars
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU84041
Record Dates: First submitted 2013-10-15; First posted 2013-11-05 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractional Radiofrequency (Active Comparator): Subjects will be randomly assigned to receive fractional radiofrequency treatment to either the right or left side of the face and the contralateral side will receive 1550-nm fractional photothermolysis. Subjects will receive treatments at baseline, week 4, and week 8 for a total of three treatments. Follow up visits will take place at week 16, two months following the last treatment visit.
  Interventions: Device: Fractional Radiofrequency
- 1550-nm Fractional Photothermolysis (Active Comparator): Subjects will be randomly assigned to receive fractional radiofrequency treatment to either the right or left side of the face and the contralateral side will receive 1550-nm fractional photothermolysis. Subjects will receive treatments at baseline, week 4, and week 8 for a total of three treatments. Follow up visits will take place at week 16, two months following the last treatment visit.
  Interventions: Device: 1550-nm Fractional Photothermolysis

INTERVENTIONS:
Device: Fractional Radiofrequency
  Other Names: ePrime
  Arms: Fractional Radiofrequency
Device: 1550-nm Fractional Photothermolysis
  Other Names: Fraxel
  Arms: 1550-nm Fractional Photothermolysis

SUMMARY:
The purpose of this study is to compare the effectiveness of the ePrime fractional radiofrequency system to the 1550-nm fractional photothermolysis system (Fraxel) in the ability to improve acne scar appearance.

DETAILED DESCRIPTION:
Participants in this study will be patients at the dermatology clinic with icepick and boxcar acne scars on at least one 2 x 2 cm area on each side of face. Subjects will be randomly assigned to receive fractional radiofrequency treatment to either the right or left side of the face and the contralateral side will receive 1550-nm fractional photothermolysis. Subjects will receive treatments at baseline, week 4, and week 8 for a total of three treatments. Follow up visits will take place at week 16, two months following the last treatment visit. This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 years and older.
2. Subjects with bilateral 2x2 cm areas of ice pick and/or boxcar acne scars on their face.
3. Subjects are in good health.
4. Subjects have the willingness and the ability to understand and provide informed consent and communicate with the investigator.

Exclusion Criteria:

1. Subjects who have received injectable soft-tissue augmentation materials to the face, or facial ablative resurfacing, within the past 6 months.
2. Subjects who have received injectable botulinum toxin to the face, or any nonablative laser treatment to the face, within the past 3 months.
3. Subjects who have local infections, open facial wounds, or other significant local skin disease that would interfere with acne scar treatment with energy devices.
4. Subjects who are allergic to lidocaine or prilocaine.
5. Subjects who have a history of abnormal scarring in the treatment area, such as keloid scar formation.
6. Subjects who have ectropion or or other eyelid disfigurement.
7. Subjects who have a history of isotretinoin use in the preceding year.
8. Pregnant or lactating individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in best overall cosmetic appearance (right side or left side better)rated by a blinded dermatologist from baseline to week 16 | 1 hour at baseline and week 16
  The primary outcome was a blinded rating of the treatment area (Fractional Radiofrequency Versus Fractional Photothermolysis) with the best cosmetic appearance. A dermatologist will blindly evaluate the treated areas of each side from live subjects at baseline and on the final follow up visit (week 16).

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States